CLINICAL TRIAL: NCT03895827
Title: Recovery Initiation and Management After Overdose (RIMO) Experiment: Phase 2 Main Clinical Trial (R33)
Brief Title: Recovery Initiation and Management After Overdose (RIMO) Experiment
Acronym: RIMO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christine Grella, Senior Research Scientist, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1132-0319; 1R21DA045774 (NIH)
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Overdose; First responders; Medication Assisted Treatment; Treatment linkage
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to experiment group getting Recovery Initiation and Management after Overdose (RIMO) intervention or control group getting a passive referral to medication assisted treatment.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is blind to the condition of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Referral Control (Active Comparator): Participants will be given information on recently expanded and publicly-funded MAT treatment in their community.
  Interventions: Other: Passive Referral to Treatment Control
- Recovery Initiation and Management after Overdose (RIMO) (Experimental): Participants assigned to the RIMO arm will meet with Linkage Managers (LM), who will use motivational interviewing (MI) techniques to: 1) identify the need for treatment and barriers to going, 2) discuss with patients the benefits of their decision to go to treatment, including activities they might enjoy as well as things they do not like about their alcohol/substance use, 3) provide personalized feedback to participants about the status of their condition based on responses to the assessment instruments, 4) help participants resolve ambivalence about their use and move them toward a commitment to change by accessing additional care, 5) address existing barriers to treatment (e.g., childcare, transportation), 6) schedule a treatment appointment, and 7) facilitate medication assisted treatment re-entry and engagement.
  Interventions: Behavioral: Recovery Initiation and Management after Overdose (RIMO); Other: Passive Referral to Treatment Control

INTERVENTIONS:
Behavioral: Recovery Initiation and Management after Overdose (RIMO) — RIMO uses motivational interviewing and linkage assistance techniques to get people who have had a recent opioid overdose reversal to go to medication-assisted treatment (MAT), stay in MAT, and, if they drop out, go back to MAT treatment.
  Arms: Recovery Initiation and Management after Overdose (RIMO)
Other: Passive Referral to Treatment Control — Currently neither first responders or emergency department staff regularly refer people to any kind of substance use after an opioid overdose reversal. In the passive referral condition they will at least get a brochure with information on recently expanded and publicly-funded medication-assisted treatment in their community.

SUMMARY:
This study targets individuals in Chicago who have received naloxone administered by first responders within the past week to reverse an overdose, but who have not entered into MAT. Study participants will be recruited through partnerships with the Chicago Fire Department (CFD) and/or Police Department (CPD); first responders will be trained to seek consent from individuals who are alert and oriented after receiving naloxone for future contacts by research staff as part of the naloxone standard protocol. Those who consent will be contacted and screened for study eligibility ideally within one week of naloxone administration; eligible participants will be randomly assigned either to the control group, i.e., referral to MAT as usual, or to Recovery Initiation and Management after Overdose (RIMO), an assertive linkage and recovery support intervention. This intervention builds on an evidence-based intervention for treatment linkage, monitoring, and recovery support evaluated in 3 prior clinical trials by the study team.

DETAILED DESCRIPTION:
Research staff will work with the Chicago Fire Department's Emergency Medical Services division and the Chicago Police Department to identify people who have just had an opioid overdose reversed with naloxone, recruit them into the trial, randomize them to a passive referral (via a brochure) vs. the RIMO experimental group. Using the study recruitment and RIMO procedures refined in Phase 1, a total of 350 individuals will be recruited and randomly assigned to the "referral to MAT" control or to "RIMO". All participants will receive standardized assessments at baseline and 3, 6, and 9 months post-randomization. The study's aims and their associated hypotheses are:

Aim 1: Evaluate RIMO's direct effect on linkage to MAT, length of time on MAT, dropout, and total days of MAT.

H1: Relative to the control group, RIMO will have a direct effect on: a) initiating MAT sooner, b) staying on medication longer, c) reducing dropout, and d) receiving more total days of MAT.

Aim 2: Evaluate RIMO's direct and indirect (via MAT) effects on time to relapse, opioid use, and opioid-related overdose.

H2: RIMO will have direct and indirect (via days of MAT treatment) effects on: a) time to relapse, b) days of opioid use, and c) number of overdoses.

Aim 3: RIMO's direct and indirect (via MAT and opioid use) effects on opioid-related fatalities, opioid use disorder (OUD) symptoms, physical health, mental health and the cost of health care utilization.

H3: RIMO will have direct and indirect (via days of MAT treatment and days of opioid use) effects on: a) opioid-related fatalities, b) opioid use disorders symptoms, c) physical health, d) mental health, and e) cost of health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* experienced an opioid overdose reversed with naloxone administered by first responders on a participating team within the past week
* not in treatment during the past 30 days
* screen positive for an OUD

Exclusion Criteria:

* under age 18
* unable to speak and understand English
* not residing in Chicago
* cognitively unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
MAT Time to Initiation | 9 months
  Days from index naloxone administration to the initiation of any kind of MAT, from treatment records.
Length of Staying on Medication | 9 months
  Days between MAT initiation and discharge, from treatment records.
MAT Days | 9 months
  Total days of MAT over 9 months from Global Appraisal of Individual Needs Quick (GAIN) and treatment records.

SECONDARY OUTCOMES:
Time to Relapse | 9 months
  Days from randomization to next subsequent use of opioids or heroin based on GAIN follow-up interviews and urine tests.
Opioid Days of Use | 9 months
  Days of opioids and/or heroin use summed over the GAIN follow-up interviews.
Opioid Overdose | 9 months
  Number of opioid-related overdose[s] summed over the GAIN follow-up interviews.
Opioid-Related Fatality | 9 months
  Any International Classification of Diseases version 10 (ICD-10) cause of death related to opioid overdose (T40.1, T40.2, T40.3, T40.4, T40.6, X42, X44, X62, X64, Y12, Y14) in Centers for Disease Control (CDC) death records.
Opioid Use Disorder symptoms | 9 months
  The Opioid Use Disorder Scale; scores range form 0 to 11 based on a count of self reported symptoms from the Diagnostic and Statistical Manual 5 criteria for opioid use disorder symptoms from the GAIN follow-up interviews. The scale score is interpreted as subclinical (0-1 symptoms), low (2-3 symptoms), moderate (4-5 symptoms) or high (6-11 symptoms) severity.
Physical Health | 9 months
  The average of 5 past 90-day items on the Health Problem Screener (worried about health, pain, health kept participant from meeting responsibilities) from GAIN follow-up interviews.
Mental Health: Internalizing Symptoms | 9 months
  The GAIN's Internalizing Disorder Screener; ranging from 0 to 6, the screener includes symptoms of depression, anxiety, trauma, suicide and are interpreted as low (0 symptoms), moderate (1-2 symptoms) or high (3-6 symptoms)
Mental Health: Externalizing Symptoms | 9 months
  The GAIN's Externalizing Disorder Screener; ranging from 0 to 6, the screener includes symptoms of attention deficit, hyperactivity, conduct, gambling disorders and are interpreted as low (0 symptoms), moderate (1-2 symptoms) or high (3-6 symptoms)
Cost of Health Care Utilization | 9 months
  Sum of the quarterly costs of health care from the GAIN-Q3 follow-up interviews; based on the frequency of health, mental health or substance-related emergency department visits, hospitalizations, residential treatment, outpatient surgery, MAT, intensive outpatient, outpatient treatment days/times multiplied by their respective costs using published estimates by health economists, adjusted for inflation using the consumer price index.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Grella, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03895827/Prot_SAP_001.pdf
  • Informed Consent Form (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03895827/ICF_000.pdf